CLINICAL TRIAL: NCT00005554
Title: Biobehavioral Predictors of Coronary Angioplasty Outcome
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5098; R29HL058638 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To examine some of the psychosocial predictors of poor outcome among revascularized coronary artery disease patients.

DETAILED DESCRIPTION:
BACKGROUND:

Percutaneous coronary revascularization procedures are increasingly used in the treatment of coronary artery disease, with approximately 300,000 interventions performed each year. Despite new developments in cardiology such as intra-coronary stents and anticoagulant pharmacological treatments, a major problem remains the frequent occurrence of coronary restenosis and new cardiac events within six months after the intervention. These adverse outcomes occur in one out of four patients and have substantial impact on the costs of medical care and patients' quality of life. Research indicated that hemostatic factors (e.g., fibrinogen, von Willebrand factor, and plasminogen activator inhibitor) promote the formation of blood clots and that these factors predict coronary restenosis. Moreover, prior longitudinal studies have also demonstrated that the psychosocial traits of hostility and depression affect clinical progression of coronary disease. These psychosocial factors significantly predict adverse long-term outcome after revascularization and both hostility and depression are known to affect blood clotting factors. In addition, acute mental and physical stress are reported to affect blood clotting factors (coagulation and fibrinolysis) and responses to stress are reported to be more pronounced in hostile individuals. However, previous research on predictors of adverse clinical outcome after percutaneous coronary revascularization has not examined stress-induced changes in hemostatic factors and the consequences of these responses for progression of coronary artery disease. Therefore, the study investigates whether psychosocial factors and responses to acute mental stress affect measures of the blood clotting process that are involved in progression of coronary disease, thereby increasing the risk of an adverse prognosis following percutaneous coronary revascularization. This study may improve the identification of patients at risk for recurrent cardiac events and provide further understanding of the pathophysiological mechanisms involved in the progression of coronary artery disease.

DESIGN NARRATIVE:

The study investigated whether psychosocial factors and responses to acute mental stress affected measures of the blood clotting process that are involved in progression of coronary disease, thereby increasing the risk of an adverse prognosis following percutaneous coronary revascularization. This study helped to improve the identification of patients at risk for recurrent cardiac events and provided further understanding of the pathophysiological mechanisms involved in the progression of coronary artery disease.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-02; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willem Kop — Uniform Services University of Health Sciences

REFERENCES:
- [Background] Kop WJ, Krantz DS, Howell RH, Ferguson MA, Papademetriou V, Lu D, Popma JJ, Quigley JF, Vernalis M, Gottdiener JS. Effects of mental stress on coronary epicardial vasomotion and flow velocity in coronary artery disease: relationship with hemodynamic stress responses. J Am Coll Cardiol. 2001 Apr;37(5):1359-66. doi: 10.1016/s0735-1097(01)01136-6. PMID 11300447
- [Background] Kop WJ, Gottdiener JS, Patterson SM, Krantz DS. Relationship between left ventricular mass and hemodynamic responses to physical and mental stress. J Psychosom Res. 2000 Jan;48(1):79-88. doi: 10.1016/s0022-3999(99)00079-3. PMID 10750633
- [Background] Kop WJ, Ader DN. Assessment and treatment of depression in coronary artery disease patients. Ital Heart J. 2001 Dec;2(12):890-4. PMID 11838334
- [Background] Kop WJ, Gottdiener JS, Tangen CM, Fried LP, McBurnie MA, Walston J, Newman A, Hirsch C, Tracy RP. Inflammation and coagulation factors in persons > 65 years of age with symptoms of depression but without evidence of myocardial ischemia. Am J Cardiol. 2002 Feb 15;89(4):419-24. doi: 10.1016/s0002-9149(01)02264-0. PMID 11835923
- [Background] Kop WJ, Verdino RJ, Gottdiener JS, O'Leary ST, Bairey Merz CN, Krantz DS. Changes in heart rate and heart rate variability before ambulatory ischemic events(1). J Am Coll Cardiol. 2001 Sep;38(3):742-9. doi: 10.1016/s0735-1097(01)01451-6. PMID 11527627
- [Background] Lundman P, Eriksson MJ, Stuhlinger M, Cooke JP, Hamsten A, Tornvall P. Mild-to-moderate hypertriglyceridemia in young men is associated with endothelial dysfunction and increased plasma concentrations of asymmetric dimethylarginine. J Am Coll Cardiol. 2001 Jul;38(1):111-6. doi: 10.1016/s0735-1097(01)01318-3. PMID 11451259
- [Background] Kop WJ. Chronic and acute psychological risk factors for clinical manifestations of coronary artery disease. Psychosom Med. 1999 Jul-Aug;61(4):476-87. doi: 10.1097/00006842-199907000-00012. PMID 10443756
- [Background] Gottdiener JS, Kop WJ, Hausner E, McCeney MK, Herrington D, Krantz DS. Effects of mental stress on flow-mediated brachial arterial dilation and influence of behavioral factors and hypercholesterolemia in subjects without cardiovascular disease. Am J Cardiol. 2003 Sep 15;92(6):687-91. doi: 10.1016/s0002-9149(03)00823-3. PMID 12972107
- [Background] Kop WJ, Vingerhoets A, Kruithof GJ, Gottdiener JS. Risk factors for myocardial infarction during vacation travel. Psychosom Med. 2003 May-Jun;65(3):396-401. doi: 10.1097/01.psy.0000046077.21273.ec. PMID 12764212
- [Background] Kop WJ, Krantz DS, Nearing BD, Gottdiener JS, Quigley JF, O'Callahan M, DelNegro AA, Friehling TD, Karasik P, Suchday S, Levine J, Verrier RL. Effects of acute mental stress and exercise on T-wave alternans in patients with implantable cardioverter defibrillators and controls. Circulation. 2004 Apr 20;109(15):1864-9. doi: 10.1161/01.CIR.0000124726.72615.60. Epub 2004 Mar 22. PMID 15037524